CLINICAL TRIAL: NCT06553976
Title: Spastic Paraplegia - Centers of Excellence Research Network (SP-CERN) - Natural History Study Pilot
Brief Title: Spastic Paraplegia - Centers of Excellence Research Network
Acronym: SP-CERN
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Columbia University (Other); University of Miami (Other); University of Michigan (Other); Baylor College of Medicine (Other); University of Texas Southwestern Medical Center (Other); University of Washington (Other); Children's Hospital Medical Center, Cincinnati (Other); Seattle Children's Hospital (Other); University of Iowa (Other)
Responsible Party: Principal Investigator, Darius Ebrahimi-Fakhari, Principal Investigator, Boston Children's Hospital
Other Study IDs: P00047458
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hereditary Spastic Paraplegia; Primary Lateral Sclerosis; SPG4; SPG5A; Spastic Paraplegia 4; Spastic Paraplegia 5A; Early Onset Hereditary Spastic Paraplegia; Neuromuscular Diseases; Spastic Paraplegia, Hereditary
MeSH Terms: conditions — Spastic Paraplegia, Hereditary; Motor Neuron Disease; Spastic Paraplegia Type 4; Neuromuscular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Spastic Paraplegia - Centers of Excellence Research Network (SP-CERN) is a collaborative research consortium dedicated to advancing the understanding, diagnosis, and treatment of hereditary spastic paraplegia (HSP) and primary lateral sclerosis (PLS). Aims of the consortium are to a) perform natural history studies of HSP subtypes, b) discover and validate biomarkers and clinician- and patient-reported outcome measures, c) uncover HSP's molecular pathophysiology and develop rational therapeutic targets, and d) perform sufficiently powered clinical trials. The current pilot study is aimed at enrolling 100 individuals with hereditary spastic paraplegia type 4 (SPG4) or hereditary spastic paraplegia type 5A (SPG5A).

DETAILED DESCRIPTION:
The hereditary spastic paraplegias (HSPs) include over 80 rare neurogenetic disorders, collectively representing the most prevalent cause of inherited spasticity and related disabilities globally. In all forms of HSP, there is a progressive deterioration of the long axonal tracts, resulting in substantial motor dysfunction and various other symptoms. Primary lateral sclerosis (PLS) is a related, degenerative neurological disorder characterized by the progressive deterioration of upper motor neurons. Both conditions result in muscle weakness and spasticity, with significant morbidity and impact on quality of life.

The Spastic Paraplegia - Centers of Excellence Research Network (SP-CERN) is a collaborative research consortium dedicated to advancing the understanding, diagnosis, and treatment of hereditary spastic paraplegia (HSP) and primary lateral sclerosis (PLS). SP-CERN provides a registry and natural history study across the whole age span, a biobank, and a genome archive. This will set the stage for a multitude of opportunities for improved diagnosis and trial readiness. A second objective is to harmonize this effort with similar consortia, especially in Europe, in addition to Asia, South America, and Africa, to help accelerate basic and clinical research on HSP and PLS on a global level. In summary, SP-CERN will support critical research infrastructure for collaborative high-quality research on HSP and PLS in North America and beyond.

General aims include:

A. Establish a shared clinical database, a repository of biospecimen samples, and a central database for the storage of all genetic data in SP-CERN.

B. Synchronize and harmonize collaborations between institutions, clinical sites, and international collaborators through the development of a central research protocol in order to standardize outcome measures and maximize the quality of research and data to ensure clinical trial readiness by regulatory standards.

C. Build comprehensive programs for advancements in diagnosis, provide more opportunities for innovative treatments, and increase access to high-quality healthcare for HSP and PLS patients.

Specific aims for this first pilot study are:

1a. Enrollment of 100 individuals with genetically-confirmed hereditary spastic paraplegia type 4 (SPG4) or hereditary spastic paraplegia type 5A (SPG5A) in the shared clinical database.

1b. Biobanking of blood samples from 100 individuals with SPG4 or SPG5A in a shared biobank.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients of all ages with a clinical and molecular diagnosis of hereditary spastic paraplegia type 4 (SPG4, SPAST) or hereditary spastic paraplegia type 5A (SPG5A, CYP7B1).

Exclusion Criteria:

* Not having such a diagnosis and/or not being related to such individual.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will enroll individuals with a known clinical and molecular diagnosis of spastic hereditary paraplegia type 4 (SPG4, SPAST) or Hereditary Spastic Paraplegia type 5A (SPG5A, CYP7B1), and/or their family members of interest (if applicable). We plan to enroll at least 100 individuals under a shared regulatory, data, and sample infrastructure over a 2-year time period.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2027-06-04 (Estimated)

PRIMARY OUTCOMES:
Establish a shared clinical database, biobank of biospecimen samples, and a central repository for the storage of all genetic data in SP-CERN. | 2 years
Synchronize collaborations between institutions and clinical sites through a central research protocol to standardize outcome measures and maximize the quality of research and data to ensure clinical trial readiness by regulatory standards. | 2 years
Test key elements in pilot projects | 2 years
Build comprehensive programs for advancements in diagnosis, provide more opportunities for innovative treatments, and increase access to high-quality healthcare for HSP and PLS patients. | 2 years

SECONDARY OUTCOMES:
Enrollment of 100 individuals with hereditary spastic paraplegia type 4 (SPG4) or hereditary spastic paraplegia type 5A (SPG5A) in the shared clinical database. | 2 years
Biobanking of blood samples from 100 individuals with SPG4 or SPG5A in a shared biobank. | 2 years

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of Iowa Carver College of Medicine, Iowa City, Iowa
  - Boston Children's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan School of Medicine, Ann Arbor, Michigan
  - Columbia University - Irving Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Scottish Rite for Children, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - University of Washington School of Medicine, Seattle, Washington

REFERENCES:
- See also: Spastic Paraplegia - Centers of Excellence Research Network Website — https://spcern.childrenshospital.org/